CLINICAL TRIAL: NCT01667887
Title: MotionLoc Study: Healing of Distal Femur Fractures Stabilized With a Flexible Plating Construct Using MotionLoc Screws
Brief Title: Plating of Distal Femur Fractures by Far Cortical Locking Using MotionLoc Screws
Status: Completed | Type: Observational
Sponsor: Legacy Biomechanics Laboratory (Other)
Collaborators: Slocum Center for Orthopedics and Sports Medicine (Other); University of Utah (Other); Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Michael Bottlang, PhD, Director, Legacy Biomechanics Laboratory, Legacy Biomechanics Laboratory
Other Study IDs: MotionLoc Screw
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Fracture of Distal Femur
Keywords: Far Cortical Locking; Distal Femur Fracture; Locking Plate; MotionLoc; Fracture Fixation
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Femur Fractures: Patients with Distal Femur Fractures

SUMMARY:
The objective of this study is to document callus formation and healing of fractures stabilized with locking plates utilizing modern MotionLoc screws that provide controlled axial micro-motion to actively promote fracture healing.

DETAILED DESCRIPTION:
Rigid locked plating constructs can suppress fracture healing, particularly at the near cortex adjacent to the plate where interfragmentary motion is minimal. Dynamic fixation with Far Cortical Locking (FCL) screws reduces construct stiffness and induces axial interfragmentary motion to stimulate symmetric callus formation and healing. Two versions of FCL screws are commercially available, but the clinical durability of this novel concept has not been documented to date. This prospective observational study documented our early clinical experience with MotionLoc® FCL screws for stabilization of distal femur fractures to assess their durability and potential complications.

Thirty-two consecutive patients with 33 distal femur fractures (AO/OTA types 33-A and 33-C) were prospectively enrolled at three trauma centers. Fractures were stabilized by plate osteosynthesis with MotionLoc® FCL screws without supplemental bone graft or bone morphogenic proteins. Thirty patients with 31 fractures were available for follow-up until union or revision. Follow-up visits at 6, 12, and 24 weeks comprised functional and radiographic assessment of implant fixation and fracture healing, including computed tomography scans at week 12. The primary endpoint was fracture healing in absence of complications and revision.

There was no incidence of implant breakage or diaphyseal fixation failure. Thirty of 31 fractures healed within 15.6 ± 6.2 weeks, as evident by bridging callus and pain-free load bearing. There were two revisions, one at 5 days post surgery to correct a mal-rotation, and one at 6 months post surgery to revise a non-union. Periosteal callus distribution at week 6 was symmetrical, with similar amounts of callus at the medial cortex (35%) anterior cortex (30%) and posterior cortex (35%). In 23 fractures (74%), callus formation extended to the lateral cortex under the plate.

Absence of hardware and fixation failure suggests that dynamic plating of distal femur fractures with FCL screws provides safe and effective fixation. Moreover, the amount and symmetric distribution of periosteal callus suggests that dynamic fixation with FCL screws may promote increased fracture healing over standard locked plating. However, this hypothesis on the stimulatory effect of dynamic fixation on fracture healing requires investigation in a future randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with distal femur fracture (AO/OTA Type 33A and 33C)
2. Patients 17 years of age and over.
3. Patients able to be operated on by selected surgeons at the participating centers.

Exclusion Criteria:

1. Pregnancy
2. Patients who are enrolled in an investigational treatment trial.
3. Patients who are not expected to survive the follow-up period.
4. Considered an inappropriate participant by the study physician.
5. Revision surgery
6. Patients currently incarcerated or awaiting incarceration.
7. Severe spinal injury with neurological deficit resulting in paralysis.
8. Fracture fixed more then 28 days after injury.
9. Acute or chronic local or systemic infections
10. Periprosthetic fractures

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Distal femur fractures (AO/OTA Type 33A and 33C)
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Fracture Healing | 6, 12, and 24 weeks post surgery
  Fracture healing is defined clinically by the ability of pain-free weight bearing, and radiographically by callus formation and bridging.

SECONDARY OUTCOMES:
Periosteal Callus Size | 6, 12, 24 weeks post surgery
  Periosteal callus size is assessed at the anterior, posterior, and medial aspects on radiographs using a validated computational algorithm.
Bridging Callus from CT | 12 weeks post surgery
  Cross-sectional image analysis, supported by 3-D rendering, to detect bony bridging at the anterior, posterior, and lateral aspects of the femur.
Fixation Failure | 24 weeks post surgery
  Assessed in terms of loss of alignment at 12 and 24 weeks post surgery
Hardware failure | 6, 12, 24 weeks post surgery
  Breakage of screw or plate

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bottlang, PhD, Principal Investigator — Legacy Biomechanics Laboratory; Steven Madey, MD, Study Chair — Legacy Health System
Locations (1):
- Legacy Health System, Portland, Oregon, United States

REFERENCES:
- See also: Orthopaedic Knowledge Online Article: Biomechanics and Use of Far Cortical Locking in Orthopaedic Trauma — http://orthoportal.aaos.org/oko/article.aspx?article=OKO_TRA041